CLINICAL TRIAL: NCT03128866
Title: Reducing Blood Loss in Hemipelvectomy Surgery With the Use Tranexamic Acid (TXA)
Brief Title: Tranexamic Acid in Reducing Blood Loss in Patients With Pelvic Tumors Undergoing Hemipelvectomy Surgery
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-0650; NCI-2018-01178 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0650 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-04-21; First posted 2017-04-25 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Pelvic Mass
MeSH Terms: interventions — Hemipelvectomy; Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (tranexamic acid) (Experimental): Patients receive tranexamic acid IV over 15 minutes 30 minutes prior to surgery and continuously during hemipelvectomy procedure in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Hemipelvectomy; Drug: Tranexamic Acid
- Arm II (no tranexamic acid) (Experimental): Patients undergo standard of care hemipelvectomy in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Hemipelvectomy

INTERVENTIONS:
Procedure: Hemipelvectomy — Undergo hemipelvectomy
Drug: Tranexamic Acid — Given IV
  Other Names: Cyclokapron; Cyklokapron; Lysteda; Tranhexamic Acid
  Arms: Arm I (tranexamic acid)

SUMMARY:
This early phase I trial studies how well tranexamic acid works in reducing the loss of blood in patients with pelvic tumors undergoing hemipelvectomy surgery. Tranexamic acid decreases blood loss by stabilizing clots and preventing clot lysis in patients undergoing surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if the use of tranexamic acid results in a significant reduction in intraoperative and perioperative blood loss.

SECONDARY OBJECTIVES:

I. To determine if use of tranexamic acid lowers the amount of blood products transfused in hemipelvectomy surgeries and during first postoperative week.

II. To determine if the use of tranexamic acid has an effect on laboratory (lab) measurements preoperatively through postoperative day 7.

III. To determine if use of tranexamic acid has an effect on complication, length of intensive care unit (ICU), and hospital stays.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (TRANEXAMIC ACID): Patients receive tranexamic acid intravenously (IV) over 15 minutes 30 minutes prior to surgery and continuously during hemipelvectomy procedure in the absence of disease progression or unacceptable toxicity.

ARM II (NO TRANEXAMIC ACID): Patients undergo standard of care hemipelvectomy in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Both pediatric and adult patients can be eligible to participate
* Cognitively impaired and non-English speakers can be eligible to participate.
* Both male and female patients must have a pelvic tumor and are scheduled to have surgery at University of Texas (UT) Monroe Dunaway (MD) Anderson Cancer center that require hemipelvectomy, resulting in pelvic ring disruption

Exclusion Criteria:

* Patient with a history of genetic prothrombotic state
* Patient with a history of thromboembolic disease to include pulmonary embolus or other extremity deep venous thrombosis
* Patients with thrombosis of the planned site of resection will not be excluded if the thrombus is caused directly by tumor burden or outflow obstruction
* Female patients will not be eligible for this study if she is either pregnant or nursing at the time of enrollment
* Patients will not be eligible if they have a history of color vision defects
* Patients will not be eligible if they have a history of retinal vein or artery occlusion
* Patients will not be eligible if they have a history of intracranial hemorrhage in past 6 months
* Patients will not be eligible if they have a history of hypersensitivity to tranexamic acid
* Patients will not be eligible if they present with moderate to severe decrease in creatinine clearance (estimated glomerular filtration rate [eGFR] < 45 mL/min/1.73m2)
* Patients will not be eligible if they present or have a history of seizure disorder

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-05-19 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Total perioperative blood loss defined as the total intraoperative estimation of blood (EBL) loss | During first post-operative week
  Intraoperative blood loss and perioperative blood loss (total of intraoperative EBL and 1 week drain) will be compared between two groups utilizing two-sample t-test or Wilcoxon rank-sum test. Log-transformation will be taken on the blood loss measurements as appropriate. Multivariable linear regression models will be used to compare two treatment groups in intraoperative and perioperative blood loss by adjusting for significant covariates. Model selection technique, including backward elimination, will be implemented.

SECONDARY OUTCOMES:
Total number of units of packed red blood cells (PRBCs), fresh frozen plasma (FFP), cryoprecipitate, and platelets | At the time of procedure
  Two groups will be compared in each of secondary outcome measures utilizing two-sample t-test or Wilcoxon rank-sum test for continuous variables (amount of blood products transfused (during operation and during first postoperative week), lab measurements, length of intense care unit (ICU), and hospital stays) and Chi-square test or Fisher's exact test for categorical variables (complication). Modeling techniques including linear regression (amount of blood products transfused, length of ICU, hospital stays), logistic regression (complication), and mixed effects model (repeatedly measured lab data) will be utilized as appropriate.
Total number of units of PRBCs, FFP, cryoprecipitate, and platelets | During first post-operative week
  Two groups will be compared in each of secondary outcome measures utilizing two-sample t-test or Wilcoxon rank-sum test for continuous variables (amount of blood products transfused (during operation and during first postoperative week), lab measurements, length of ICU, and hospital stays) and Chi-square test or Fisher's exact test for categorical variables (complication). Modeling techniques including linear regression (amount of blood products transfused, length of ICU, hospital stays), logistic regression (complication), and mixed effects model (repeatedly measured lab data) will be utilized as appropriate.
Thromboelastography (TEG) | At baseline prior to administration of tranexamic acid, after completion of bone cuts, and after completion of closure
  Two groups will be compared in each of secondary outcome measures utilizing two-sample t-test or Wilcoxon rank-sum test for continuous variables (amount of blood products transfused (during operation and during first postoperative week), lab measurements, length of ICU, and hospital stays) and Chi-square test or Fisher's exact test for categorical variables (complication). Modeling techniques including linear regression (amount of blood products transfused, length of ICU, hospital stays), logistic regression (complication), and mixed effects model (repeatedly measured lab data) will be utilized as appropriate.
Change in laboratory measurements | Baseline up to 7 days post-surgery
  Two groups will be compared in each of secondary outcome measures utilizing two-sample t-test or Wilcoxon rank-sum test for continuous variables (amount of blood products transfused (during operation and during first postoperative week), lab measurements, length of ICU, and hospital stays) and Chi-square test or Fisher's exact test for categorical variables (complication). Modeling techniques including linear regression (amount of blood products transfused, length of ICU, hospital stays), logistic regression (complication), and mixed effects model (repeatedly measured lab data) will be utilized as appropriate.
Complications including but not limited to venous thromboembolism, stroke, seizure, vision changes, and return to operating room (hematoma, active bleeding) | Up to 7 days post-surgery
  Two groups will be compared in each of secondary outcome measures utilizing two-sample t-test or Wilcoxon rank-sum test for continuous variables (amount of blood products transfused (during operation and during first postoperative week), lab measurements, length of ICU, and hospital stays) and Chi-square test or Fisher's exact test for categorical variables (complication). Modeling techniques including linear regression (amount of blood products transfused, length of ICU, hospital stays), logistic regression (complication), and mixed effects model (repeatedly measured lab data) will be utilized as appropriate.
Length of ICU and hospital stay | Up to 7 days post-surgery
  Two groups will be compared in each of secondary outcome measures utilizing two-sample t-test or Wilcoxon rank-sum test for continuous variables (amount of blood products transfused (during operation and during first postoperative week), lab measurements, length of ICU, and hospital stays) and Chi-square test or Fisher's exact test for categorical variables (complication). Modeling techniques including linear regression (amount of blood products transfused, length of ICU, hospital stays), logistic regression (complication), and mixed effects model (repeatedly measured lab data) will be utilized as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Valerae O Lewis, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org